CLINICAL TRIAL: NCT00069030
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of the HIV-1 DNA Vaccine VRC-HIVDNA009-00-VP (Gag-Pol-Nef-multiclade Env) With the Plasmid Cytokine Adjuvant VRC-ADJDNA004-IL2-VP (IL-2/Ig)
Brief Title: Safety of and Immune Response to an HIV Vaccine (VRC-HIVDNA009-00-VP) Administered With Interleukin-2/Immunoglobulin (IL-2/Ig) DNA Adjuvant in Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 044; 5K08AI051223-03 (NIH); 10120 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2003-09-12; First posted 2003-09-16 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; HIV-1; AIDS Vaccines; Vaccines, DNA; Dose-Response Relationship, Immunologic; Cytokines; Plasmids; Adjuvants, Immunologic; Drug Administration Schedule; Interleukin; IL2; Ig; IL@/Ig
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: VRC-HIVDNA009-00-VP (Gag-Pol-Nef-multiclade-Env) with adjuvant VRC-ADJDNA004-IL2-VP

SUMMARY:
This study will test the safety of and immune system response to a new HIV vaccine. The vaccine in this study is made from HIV DNA produced in a laboratory. Only part of the virus's DNA is used in the vaccine and the vaccine itself cannot cause HIV infection or AIDS. In addition to HIV DNA, the vaccine contains interleukin-2 (IL-2) DNA fused to a portion of immunoglobulin (Ig) DNA. IL-2 is a chemical that stimulates the immune system and may improve response to the vaccine.

Study hypothesis: The IL-2/Ig plasmid will be very well tolerated in humans.

DETAILED DESCRIPTION:
Over 90% of the 40 million people infected with HIV live in developing countries and have little or no access to antiretroviral medications. The worldwide HIV/AIDS epidemic will only be controlled through development of a safe and effective vaccine that will prevent HIV infection. DNA vaccines are inexpensive to construct, readily produced in large quantities, and stable for long periods of time. The DNA vaccine in this study, VRC-HIVDNA009-00-VP (Gag-Pol-Nef-multiclade Env), uses multiple gene products to increase the breadth of the immune response across different HIV subtypes. The DNA plasmids in VRC-HIVDNA009-00-VP code for proteins from HIV subtypes A, B, and C, which together represent 90% of new HIV infections in the world.

The study vaccine is administered with an adjuvant. The adjuvant is a DNA plasmid encoding interleukin 2 (IL-2) fused to the Fc portion of IgG for enhanced stability. This IL-2/Ig adjuvant may augment the immune system's response to the vaccine.

Participants in this study will be randomly assigned to receive either the vaccine and adjuvant, the vaccine and placebo, the adjuvant and placebo, or placebo alone. All injections will be administered by needle-free injection in the upper arm. Participants will receive four does of vaccine: one at their first study visit and then at Months 1, 2, and 6. Participants will have a follow-up visit 2 days after each injection. Some participants may receive another injection at this follow-up visit. All study participants will be followed for 18 months and will have 16 to 20 study visits. Study visits will last 1/2 to 2 hours and will include blood and urine tests and a physical exam. Participants will also have six HIV tests over the course of the study.

ELIGIBILITY:
Inclusion Criteria

* HIV negative
* Willing to receive HIV test results
* Good general health
* Acceptable methods of contraception for females of reproductive potential
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV is positive
* Normal thyroid stimulating hormone (TSH) level

Exclusion Criteria

* HIV vaccines or placebos in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Clinical depression with pharmacological treatment within the past 2 years
* Active syphilis
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Unstable asthma
* Type 1 or Type 2 Diabetes Mellitus
* Thyroid disease requiring treatment
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgement of the investigator, would interfere with the study
* Pregnant or breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2003-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Clinical observation and monitoring of hematological, chemical, and immunologic parameters
local and systemic adverse reactions after each injection and for 12 months after last injection

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Dolin, MD, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (7):
- United States (7):
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - NY Blood Ctr./Union Square CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island

REFERENCES:
- [Background] Barouch DH, Santra S, Schmitz JE, Kuroda MJ, Fu TM, Wagner W, Bilska M, Craiu A, Zheng XX, Krivulka GR, Beaudry K, Lifton MA, Nickerson CE, Trigona WL, Punt K, Freed DC, Guan L, Dubey S, Casimiro D, Simon A, Davies ME, Chastain M, Strom TB, Gelman RS, Montefiori DC, Lewis MG, Emini EA, Shiver JW, Letvin NL. Control of viremia and prevention of clinical AIDS in rhesus monkeys by cytokine-augmented DNA vaccination. Science. 2000 Oct 20;290(5491):486-92. doi: 10.1126/science.290.5491.486. PMID 11039923
- [Background] Barouch DH, Santra S, Steenbeke TD, Zheng XX, Perry HC, Davies ME, Freed DC, Craiu A, Strom TB, Shiver JW, Letvin NL. Augmentation and suppression of immune responses to an HIV-1 DNA vaccine by plasmid cytokine/Ig administration. J Immunol. 1998 Aug 15;161(4):1875-82. PMID 9712056
- [Background] Moore JP, Parren PW, Burton DR. Genetic subtypes, humoral immunity, and human immunodeficiency virus type 1 vaccine development. J Virol. 2001 Jul;75(13):5721-9. doi: 10.1128/JVI.75.13.5721-5729.2001. No abstract available. PMID 11390574
- [Background] Approaches to the development of broadly protective HIV vaccines: challenges posed by the genetic, biological and antigenic variability of HIV-1: Report from a meeting of the WHO-UNAIDS Vaccine Advisory Committee Geneva, 21-23 February 2000. AIDS. 2001 Apr 13;15(6):W1-W25. No abstract available. PMID 11371709
- [Background] Walker LG, Walker MB, Heys SD, Lolley J, Wesnes K, Eremin O. The psychological and psychiatric effects of rIL-2 therapy: a controlled clinical trial. Psychooncology. 1997 Dec;6(4):290-301. doi: 10.1002/(SICI)1099-1611(199712)6:43.0.CO;2-G. PMID 9451748
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067
- [Derived] Baden LR, Blattner WA, Morgan C, Huang Y, Defawe OD, Sobieszczyk ME, Kochar N, Tomaras GD, McElrath MJ, Russell N, Brandariz K, Cardinali M, Graham BS, Barouch DH, Dolin R; NIAID HIV Vaccine Trials Network 044 Study Team. Timing of plasmid cytokine (IL-2/Ig) administration affects HIV-1 vaccine immunogenicity in HIV-seronegative subjects. J Infect Dis. 2011 Nov 15;204(10):1541-9. doi: 10.1093/infdis/jir615. Epub 2011 Sep 21. PMID 21940420